CLINICAL TRIAL: NCT03440944
Title: Superior Venous Access, Midline vs Ultrasound IVs: A Randomized Clinical Trial
Brief Title: Superior Venous Access, Midline vs Ultrasound IVs
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was stopped after a pause due to COVID-19 policies and new published evidence about the effectiveness of the interventon.
Sponsor: Boston Medical Center (Other)
Collaborators: Society for Academic Emergency Medicine (Other); Bard Peripheral Vascular, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-37285; H-37285 (Other Grant/Funding Number: Society for Academic Emergency Medicine); H-37285 (Other Grant/Funding Number: Bard Peripheral Vascular, Inc.)
Record Dates: First submitted 2018-01-11; First posted 2018-02-22 (Actual); Results first posted 2021-04-29 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Vascular Access Complication; Ultrasound Therapy; Complications
Keywords: vascular access; midline cather; ultrasound guided IV

STUDY DESIGN:
Intervention Model Description: randomized to one of two therapies, peripheral ultrasound IV or midline
Masking Description: Given the devices are different we will not be able to mask.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Ultrasound Guided Peripheral IV Catheter (Active Comparator): Patients if randomized to this group will receive a standard ultrasound guided peripheral IV. The IV is 4.88cm in length.
  Interventions: Device: Ultrasound Guided Peripheral IV Catheter
- Midline Catheter (Active Comparator): Patients if randomized to this group will receive a midline catheter. The catheter is 10cm in length.
  Interventions: Device: Midline Catheter

INTERVENTIONS:
Device: Ultrasound Guided Peripheral IV Catheter — Patients randomized to this arm will receive an ultrasound guided peripheral IV catheter.
  Arms: Ultrasound Guided Peripheral IV Catheter
Device: Midline Catheter — Patients randomized to this group will receive a midline catheter. The catheter is 10cm in length.
  Arms: Midline Catheter

SUMMARY:
Obtaining intravenous access (IVA) is the most common procedure performed in the emergency department (ED). Placement of IVA allows for blood work and delivery of intravenous fluids and medications. The implementation of ultrasound guided peripheral IVs (UGPIV) have allowed for ultrasound to be used to place an IV into patients with difficult vein access (DVA). An alternative device to place is a midline catheter (MC). The use of MCs against UGPIV has not been compared in a randomized study. Aim 1: To determine if UGPIVs have a higher failure rate than midline catheters within 72 hours of placement. Aim 2: To collect information to perform a direct cost analysis of UGPIV against that of the midline catheter. Aim 3: Assess patient satisfaction.

DETAILED DESCRIPTION:
This is a randomized controlled trial to determine if the midline catheter is superior to the ultrasound guided IV with respect to survival at 72 hours.

Aim 1: To determine if UGPIVs have a higher failure rate than midline catheters within 72 hours of placement. There are several reasons why UGPIVs may fail. UGPIVs are shorter than midline catheters, and shorter catheters may fail due to infiltration which can be a result of malposition as well as having the catheter pull out of the vessel. It is being hypothesized that by using a midline catheter with a guidewire for placement with additional catheter length placed into the vessel, midlines will be superior to UGP\Vs with regards to survival time of the catheter. The investigators will assess catheter survival daily until 72 hours (when UGPIV are recommended to be changed). The total lifetime of the midline catheters will be recorded.

Aim 2: To perform a direct cost analysis of UGPIV against that of the midline catheter. This study will not be large enough to complete a robust cost effectiveness analysis to compare UGPIV to mid line catheters. As a part of this study the investigators will collect information including but not limited to: the number of catheters used for IVA attempts, time for placement of each device complications, and need for additional IVA during hospitalization.

Aim 3: For patients that remain hospitalized at 72 hours a satisfaction survey will be administered to determine patient experience and preference for the type of vascular access that they receive.

ELIGIBILITY:
Inclusion Criteria:

* Patient at least 18 years of age being treated in the emergency department at Boston Medical Center
* Standard IVA cannot be obtained by two qualified ER staff
* Have an upper extremity (left or right arm) that can accept a deep venous IV
* Clinical team believes the patient is likely to require inpatient admission at time of needing IV access
* English speaking
* Able to provide consent

Exclusion Criteria:

* Patient expected to be discharged from the emergency department or discharged from the hospital within 1 nights stay.
* Prisoner
* Pregnancy
* Requires central line or midline catheter as an expected requirement of care
* Patients who are expected to require medication that is not approved for administration via a peripherally guided IV or midline as defined by hospital pharmacy guidelines.
* Patients known to have bacteremia or have a high suspicion of bacteremia
* The patient is known or is suspected to be allergic to materials contained in the device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-04-23 (Actual); Primary Completion 2021-01-25 (Actual); Study Completion 2021-01-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Pare, MD MHS RDMS, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tada M, Yamada N, Matsumoto T, Takeda C, Furukawa TA, Watanabe N. Ultrasound guidance versus landmark method for peripheral venous cannulation in adults. Cochrane Database Syst Rev. 2022 Dec 12;12(12):CD013434. doi: 10.1002/14651858.CD013434.pub2. PMID 36507736

RESULTS

PARTICIPANT FLOW:
Groups:
- Ultrasound Guided Peripheral IV Catheter: Patients if randomized to this group will receive a standard ultrasound guided peripheral IV. The IV is 4.77cm in length.
  Ultrasound Guided Peripheral IV Catheter: Patients randomized to this arm will receive an ultrasound guided peripheral IV catheter.
Period: Overall Study
Arm/Group | Ultrasound Guided Peripheral IV Catheter | Midline Catheter
Started | 9 | 9
Completed | 8 | 8
Not Completed | 1 | 1
Not completed — Physician Decision | 1 | 0
Not completed — No Acceptable Vasculature | 0 | 1

BASELINE CHARACTERISTICS:
Population: Only patients that received Ultrasound Guided Peripheral IV or Midline Catheter underwent analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ultrasound Guided Peripheral IV Catheter | Midline Catheter | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 7 | 14
  >=65 years | 1 | 1 | 2
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 42 [36 to 58] | 53 [43 to 62] | 49 [38 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 2 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 8 | 6 | 14
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 5 | 10
  White | 3 | 3 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: Device Failures Within 72 Hours
Description: Total number and percentage of device failures within 72 hours of placement based on midline and ultrasound guided peripheral IV catheter. Medical record review and in person visits with medical treatment teams and patients were used to assess if device failure occurred within 72 hours. Device failure was determined by needing to have any device replaced or removed for clinical care.
Time Frame: 72 hours after device placement
Population: Patients who completed therapy within 72 hours were considered non-failure
Measure: Count of Participants; unit: Participants
Arm/Group | Ultrasound Guided Peripheral IV Catheter | Midline Catheter
Number analyzed (Participants) | 8 | 8
Participants
  Device Failure within 72 hours | 6 | 1
  No Device Failure within 72 hours | 2 | 7

2. Secondary Outcome: IV Catheter Insertion Time
Description: The time it takes to insert the IV catheter will be documented in minutes for each study participant.
Time Frame: from catheter insertion
Population: Time taken to place each device
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Ultrasound Guided Peripheral IV Catheter | Midline Catheter
Number analyzed (Participants) | 8 | 8
minutes | 9 [7 to 13] | 17.5 [14 to 25]

3. Secondary Outcome: Total Number of Replacement Catheters
Description: The total number of replacement IV catheters will be documented. This will be assessed based on each group (Ultrasound Guided Peripheral IV Catheter and Midline Catheter).
Time Frame: from catheter insertion up to 30 days
Population: Number of additional IV (including Midline) catheters placed
Measure: Number; unit: additional IV access devices
Arm/Group | Ultrasound Guided Peripheral IV Catheter | Midline Catheter
Number analyzed (Participants) | 8 | 8
additional IV access devices | 13 | 1

4. Secondary Outcome: Catheter Related Costs
Description: The mean costs per patient associated with the placement and replacement of catheters for each participant will be calculated.
Time Frame: from catheter insertion up to 30 days
Measure: Mean (Standard Deviation); unit: US Dollars
Arm/Group | Ultrasound Guided Peripheral IV Catheter | Midline Catheter
Number analyzed (Participants) | 8 | 8
US Dollars | 38.25 (21.95) | 28.88 (4.68)

5. Secondary Outcome: Patient Satisfaction
Description: Participant experience and satisfaction will be assessed with a short survey that will be given to participants who stay at least 72 hours after catheter insertion.
Time Frame: 72 hours after catheter insertion
Population: Patients who stayed for 72 hours, preference to have midline over ultrasound guided peripheral IV catheter. Patients discharged prior to 72 hours of therapy are not included in the reported results. For the Midline Catheter arm only 3 participants stayed at least 72 hours; 5 participants did not complete the satisfaction survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Ultrasound Guided Peripheral IV Catheter | Midline Catheter
Number analyzed (Participants) | 8 | 3
Participants
  Prefer Midline | 4 | 3
  Unsure | 3 | 0
  No | 1 | 0

ADVERSE EVENTS:
Time Frame: Within 30 days of IV or Midline device placement
Description: Adverse Event included device failure or required replacement.
Arm/Group | Ultrasound Guided Peripheral IV Catheter | Midline Catheter
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 6/8 | 1/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ultrasound Guided Peripheral IV Catheter (N=8) | Midline Catheter (N=8)
Device Failure (Surgical and medical procedures) | 6 (6) | 1 (1) — Device failure due to either pain, swelling, being dislodged, infiltration, or other failure such as inability to provide medications.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-29): https://cdn.clinicaltrials.gov/large-docs/44/NCT03440944/Prot_SAP_000.pdf